CLINICAL TRIAL: NCT01031420
Title: Phase II Trial of Neoadjuvant Dose Dense MVAC in Muscle Invasive Bladder Cancer and High Risk Urothelial Carcinoma of the Upper Urinary Tract
Brief Title: Dose Dense MVAC for Muscle Invasive Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FER-GU-026; NCI-2010-01910 (Registry Identifier: NCI Clinical Trials Reporting Office)
Record Dates: First submitted 2009-12-03; First posted 2009-12-14 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-08

CONDITIONS: Muscle Invasive Bladder Cancer; High Risk Urothelial Carcinoma of the Upper Urinary Tracts
Keywords: bladder; cancer; invasive
MeSH Terms: conditions — Neoplasms | interventions — Methotrexate; Sodium; merphos; Vinblastine; Doxorubicin; Cisplatin; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dose dense MVAC (Experimental): standard doses of MVAC given every 14 days x 3.
  Interventions: Drug: single arm dose dense MVAC

INTERVENTIONS:
Drug: single arm dose dense MVAC — standard doses of methotrexate, vinblastine, adriamycin, and cisplatin given every 14 days.
  Other Names: methotrexate (MTX) sodium; MTX; Mexate; Mexate-AQ; Foex; Folex; Abitrexate; Rheumatrex; amethopterin; Velban; Velsar; AlkabanAQ; Velbe; vinblastine sulfate; vincaleukoblastine; VLB; doxorubicin; doxorubicin hydrochloride liposomal Doxil,; Rubex; Adria; cis-platinum, cisdiammineddichloroplatinum,; CDDP; Platinol; platinum

SUMMARY:
Standard treatment for early stage bladder cancer is chemotherapy with methotrexate (M), vinblastine (V), adriamycin (A), and cisplatin (C) followed by surgical removal of any remaining cancer and the bladder with the intent of cure. The M V chemotherapy is usually given every 14 days with the AC given along each 28 days. This study looks at giving the same drugs at the same doses closer together, all drugs every 14 days, with the support of growth factor medication to promote growth of the white blood cells and platelets and allow chemotherapy to be finished sooner and surgery to be done sooner.

DETAILED DESCRIPTION:
Primary Objective To assess the rate of complete response (pT0) at cystectomy or ureterectomy following preoperative dose dense MVAC (DD-MVAC) in patients with muscle invasive urothelial carcinoma of the bladder or high grade upper tract urothelial carcinoma.

Secondary Objectives To assess the toxicity profile of DD-MVAC when given in the neoadjuvant setting: To define the number of patients who complete all three cycles of treatment without dose reduction, and to compare incidence of toxicity to the historical standard described by Grossman et al. To assess the 5 year overall and relapse free survival in patients who receive neoadjuvant DD-MVAC. To compare complete response rates between the following subgroups of study patients: Among bladder patients: Clinical N0 versus N1 (Appendix B) Among bladder patients: T2 stage without high risk features versus T2 with high risk features plus those with > T2 stage.

Three 14 day cycles of:

Methotrexate 30 mg/m2 IV push or infusion over 2-3 minutes. Day 1

Vinblastine 3 mg/m2 Slow IV push or infusion over Day 1

Doxorubicin 30 mg/m2 Slow IV push or infusion over 15 minutes Day 1

Cisplatin 70 mg/m2 IV infusion over 4 hours Note: May divide dose over two sequential days (35 mg/m2/d x 2 days) if creatinine clearance 50-59 mL/min Day 1* (or divided over Day 1 and Day 2)

Pegfilgrastim 6 mg subcutaneous (SQ) 24-48 hours after completion of chemotherapy.

Followed in 4-8 weeks by radical cystectomy/ureterectomy.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed urothelial carcinoma of bladder, ureter, or renal pelvis. T2-T4 and muscle invasion must be established by TURBT. Upper tract must be high grade. N0-N1 are eligible.
* candidate for radical cystectomy, nephroureterectomy, or segmental ureterectomy with goal of cure.

  ->/= 18 years old
* ECOG performance status 0-1.
* Adequate marrow and organ function.
* May enter on therapeutic anticoagulation if it can be safely held during perioperative period.
* No women of childbearing potential, pregnant or breastfeeding.
* LVEF >/= 50 %
* Patients with history of other non-urothelial malignancies may enroll if: 1)no evidence of distant disease w/in last year. 2)No anticancer treatment for >/= 1 year other than adjuvant treatment or treatment for secondary prevention. 3) Less than 360 mg/m2 lifetime dose of adriamycin.
* ability to understand and willingness to sign written informed consent and HIPAA.

Exclusion Criteria:

* Intravesicular therapy w/in 4 weeks of study entry or those who have not recovered from adverse effects of such agents administered more than 4 weeks earlier.
* Patients may not be receiving any investigational agents within 4 weeks of study entry.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Methotrexate, Vinblastine, Adriamycin or Cisplatin or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study due to the potential for teratogenic or abortifacient effects of cytotoxic chemotherapy.
* Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with cytotoxic chemotherapy. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.

  -. Patients who have undergone prior pelvic radiation are excluded due to risk of life threatening myelosuppression.
* Patients who have received any previous systemic chemotherapy or radiation therapy for urothelial carcinoma or cytotoxic chemotherapy for another malignancy within 1 year of study entry are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-12-07 (Actual); Primary Completion 2013-07-19 (Actual); Study Completion 2013-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Plimack, MD, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Plimack ER, Hoffman-Censits JH, Viterbo R, Trabulsi EJ, Ross EA, Greenberg RE, Chen DY, Lallas CD, Wong YN, Lin J, Kutikov A, Dotan E, Brennan TA, Palma N, Dulaimi E, Mehrazin R, Boorjian SA, Kelly WK, Uzzo RG, Hudes GR. Accelerated methotrexate, vinblastine, doxorubicin, and cisplatin is safe, effective, and efficient neoadjuvant treatment for muscle-invasive bladder cancer: results of a multicenter phase II study with molecular correlates of response and toxicity. J Clin Oncol. 2014 Jun 20;32(18):1895-901. doi: 10.1200/JCO.2013.53.2465. Epub 2014 May 12. PMID 24821881
- See also: Pubmed.gov — http://www.ncbi.nlm.nih.gov/pubmed/?term=24821881

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Dense MVAC
Started | 54
Completed | 44
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Dose Dense MVAC
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 28
Age, Continuous [Median (Full Range); unit: years] | 65 [44 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response at Cystectomy or Ureterectomy Following Preoperative Dose Dense MVAC
Description: complete response rate (pT0), as defined by pathologic staging at cystectomy or ureterectomy, following neoadjuvant DD-MVAC chemotherapy.
Time Frame: Following completion of the 3rd/final cycle of chemotherapy (about week 9) by CT imaging and at time of surgery for pathologic response.
Measure: Number (95% Confidence Interval); unit: percentage of total participants
Arm/Group | Dose Dense MVAC
Number analyzed (Participants) | 44
percentage of total participants | 38 [23 to 53]

2. Secondary Outcome: Toxicity Profile of Dose Dense MVAC Given in the Neoadjuvant Setting.
Description: Defined by number of patients who complete all three cycles of treatment without dose reduction
Time Frame: Ongoing throughout treatment at each MD visit every 14 days.
Population: Forty patients were evaluable for response as predefined in the protocol.
Measure: Number; unit: participants
Arm/Group | Dose Dense MVAC
Number analyzed (Participants) | 40
participants
  All three cycles of chemotherapy were completed | 37
  Discontinued chemotherapy | 3

ADVERSE EVENTS:
Arm/Group | Dose Dense MVAC
Serious Adverse Events (participants affected / at risk) | 22/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Dense MVAC (N=40)
Anemia (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 3
Lymphocytopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Sepsis (Infections and infestations) | 1
proteinuria (Renal and urinary disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Pharyngitis (Infections and infestations) | 1
Mucositis (Gastrointestinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
hypokalemia (Metabolism and nutrition disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
hyperkalemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No